CLINICAL TRIAL: NCT00618709
Title: Phase 1, Open-Label, Dose-Escalation Safety and Pharmacokinetic Study of ATX-101 (Sodium Deoxycholate for Injection) Following Subcutaneous Injections in the Submental Area
Brief Title: Dose-Escalation Safety and Pharmacokinetic Study of ATX-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ATX-101-07-08; ATX-101-07-08
Record Dates: First submitted 2008-01-23; First posted 2008-02-20 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): ATX-101 (1 mg/cm2) at a volume of 0.2 ml on a 1.0 cm grid
  Interventions: Drug: ATX-101
- Cohort 2 (Experimental): ATX-101 (2 mg/cm2) at a volume of 0.2 ml on a 1.0 cm grid
  Interventions: Drug: ATX-101
- Cohort 3 (Experimental): 3 subgroups in Cohort 3: 3a: ATX-101 (4 mg/cm2) at a volume of 0.2 ml on a 1.0 cm grid 3b: ATX-101 (2 mg/cm2) at a volume of 0.2 ml on a 0.7 cm grid 3c: ATX-101 (2 mg/cm2) at a volume of 0.4 ml on a 1.0 cm grid
  Interventions: Drug: ATX-101
- Cohort 4 (Experimental): 3 subgroups in Cohort 4: 4a: ATX-101 (8 mg/cm2) at a volume of 0.2 ml on a 1.0 cm grid 4b: ATX-101 (4 mg/cm2) at a volume of 0.2 ml on a 0.7 cm grid 4c: ATX-101 (4 mg/cm2) at a volume of 0.4 ml on a 1.0 cm grid
  Interventions: Drug: ATX-101

INTERVENTIONS:
Drug: ATX-101 — ATX-101 single dose

SUMMARY:
The purpose of this research is to evaluate the safety and pharmacokinetic profile of single doses of ATX-101

DETAILED DESCRIPTION:
This is a single center, open-label, dose-escalation study in which subjects will receive 4 different dosage concentrations (3 dosing paradigms) of ATX-101 in a single dosing session.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or nonpregnant females
* Age 18 to 65
* Sufficient submental fat for injections
* Signed informed consent

Exclusion Criteria:

* Prior interventions in the chin or neck area
* History or presence of drug or alcohol abuse
* Treatment with an investigational agent within 30 days before the dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety assessed by: Laboratory tests | 12 weeks
Safety assessed by: medical evaluations | 24 weeks
Safety assessed by: ECG results | 24 weeks

SECONDARY OUTCOMES:
Pharmacokinetic profile | 24 hours, before and after dosing
  Cmax, tmax, AUC

OTHER OUTCOMES:
Pain assessed by visual analog scale | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Swearingin, M.D., Principal Investigator — MDS Pharma Services; Frederick Beddingfield, M.D., Study Director — Sponsor GmbH
Locations (1):
- MDS Pharma Services, Tempe, Arizona, United States